CLINICAL TRIAL: NCT05596513
Title: Effectiveness of Intensive Motor Learning Approaches From Working on a Vertical Surface on Hemiplegic Children's Upper Limb Motor Skills
Brief Title: Motor Learning Approaches From Working on a Vertical Surface in Hemiplegic Children's Upper Limb Motor Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omnya Samy Abdallah Ghoneim (Other)
Responsible Party: Sponsor-Investigator, Omnya Samy Abdallah Ghoneim, Lecturer, Department of Physical Therapy for Pediatrics and Pediatric Surgery, Faculty of Physical Therapy, Badr University in Cairo, Egypt., Badr University
Organization: Badr University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003981
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Hemiplegia; Spastic
Keywords: motor learning; vertical surface; hemiplegia; cerebral palsy
MeSH Terms: conditions — Hemiplegia; Muscle Spasticity; Cerebral Palsy | interventions — Occupational Therapy

STUDY DESIGN:
Intervention Model Description: received the intensive motor-learning approaches that focuses on training of the affected hand (motor-learning approaches such as - constraint-induced movement therapy (CIMT) and hand-arm bimanual intensive training (HABIT) of the control group but from a vertical surface
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): received intensive motor-learning approaches that focuses on training of the affected hand (motor-learning approaches such as - constraint-induced movement therapy (CIMT) and hand-arm bimanual intensive training (HABIT) provide an alternative).
  Interventions: Other: motor learning and occupational therapy
- study group (Experimental): received the intensive motor-learning approaches of the control group but from a vertical surface
  Interventions: Other: Motor Learning Approaches From Working on a Vertical Surface

INTERVENTIONS:
Other: motor learning and occupational therapy — 1. Constraint-induced movement therapy (CIMT)
  2. Hand-arm bimanual intensive training (HABIT)
  Arms: control group
Other: Motor Learning Approaches From Working on a Vertical Surface — 1. Ball on wall, kneel to stand
  2. Kneel walk cross over
  3. Vertical playground puzzles and games
  4. Color on big boxes
  5. Fridge magnets
  6. Erasing a whiteboard or chalkboard
  7. Tactile feedback from textured walls
  Arms: study group

SUMMARY:
Working on a vertical surface is one of the best activities children can do to make themselves more successful in many areas as an infant which builds all those foundational skills required for the all-important task of handwriting.

DETAILED DESCRIPTION:
Motor-learning approaches such as - constraint-induced movement therapy (CIMT) offer an array of sensorimotor experiences in a playful yet repetitive and intense fashion.

A stable shoulder girdle is the co-contraction of muscles around the scapula and shoulder joint.

Depending on the activity, vertical surfaces will have kids moving their arms frequently; reaching up, down, out and around. This supports extension of the arm and an opportunity to strengthen those muscles.

Vertical surfaces facilitate wrist extension. When the wrist is extended, the ring and pinky finger tend to naturally find their way into the palm creating a more optimal grasp pattern. A child is going to be able to execute more precise and legible work when using a functional tripod or quadrupod grasp.

ELIGIBILITY:
Inclusion Criteria:

1. Children diagnosed with spastic hemiplegic cerebral palsy
2. Age 5 to 9 years
3. Manual Ability Classification System (MACS)19 scores I, II.
4. Children who can understand and cooperate with researcher's instructions
5. Children with no visual or hearing impairment

Exclusion Criteria:

1. Children with any surgical interference in the upper limb.
2. Intellectual disability such that simple tasks could not be understood or executed.
3. Inability to combine the study protocol with the regular school program

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
QUEST | 3 month
  quality of upper extremity skills test (Only dissociated movement, grasp and weight bearing domains QUEST will be assessed).

CONTACTS AND LOCATIONS:
Overall Officials: Omnya samy, PHD, Principal Investigator — lecturer
Locations (1):
- Badr University, Badr, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
individual participant data is a private data for this research